CLINICAL TRIAL: NCT03799471
Title: Somatosensory Profiles in Individuals With Persistent Musculoskeletal Pain and Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of Otago (Other)
Responsible Party: Principal Investigator, Corey Siegel, Section Chief, Gastroenterology and Hepatology, Dartmouth-Hitchcock Medical Center
Other Study IDs: W19040
Record Dates: First submitted 2019-01-06; First posted 2019-01-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Diseases; Chronic Pain; Central Sensitization
Keywords: chronic musculoskeletal pain; central hypersensitivity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD with MSK pain: IBD patients with self-reported MSK pain. No intervention. Participants will be assessed once regarding: somatosensory functioning, psychological features, MSK pain features, co-morbidity, and IBD features
- IBD without MSK pain: IBD patients without self-reported MSK pain. No intervention. Participants will be assessed once regarding: somatosensory functioning, psychological features, co-morbidity, and IBD features
- Healthy Controls: Healthy controls. No intervention. Participants will be assessed once regarding: somatosensory functioning, psychological features, and co-morbidity.

SUMMARY:
This study evaluates nervous system hypersensitivity in individuals with inflammatory bowel disease (IBD) and experiences of ongoing musculoskeletal (MSK) pain. Previous results and current literature suggest that MSK pain in IBD may be influenced by hypersensitivity of the central nervous system, termed central sensitization. However, specific mechanisms contributing to pain experiences are unknown. Therefore, primary aims are to explore aspects of central sensitization through sensory testing in this population, and to investigate association of psychological and IBD features to sensory profiles. This study hypothesizes that IBD patients with MSK pain will demonstrate altered sensory function, and IBD/psychosocial features will be associated with altered sensory functioning and worse pain experiences.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* Clinical diagnosis of IBD or healthy control

Exclusion Criteria: Participants with IBD (with and without MSK pain) will be excluded if they report any of the following:

* pregnancy
* current history of drug or alcohol abuse
* any condition resulting in altered sensation such as: nerve injuries, neurological conditions (e.g. stroke, multiple sclerosis, and Parkinson's disease)
* surgery within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dartmouth-Hitchcock Medical Center - IBD Center patient database.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold (PPT) | Baseline
  PPT will be assessed using an electronic handheld algometer (Wagner Force One™ FDIX) in: 1) low back (local), and 2) contralateral tibialis anterior. Individuals in "IBD with MSK pain" group will undergo an additional PPT assessment related to the region identified as their "main" area of MSK pain.
  PPT will be assessed by a series of 3 ascending stimulus intensities given as a slowly increasing ramp (50 kilopascal (kPa/s)) from 0 to a maximum pressure of 1000 kPa. Pressure corresponding to the moment when participants identify that the sensation of pressure alone changing to one of pressure and pain, will be recorded for each trial. PPT for each region will be described as the mean of three trials in kPa. Decreased values indicates hypersensitivity of the nervous system.
Conditioned pain modulation (CPM) | Baseline
  CPM in the present study includes: PPT of tibialis anterior (test stimulus) and cold pressor test (CPT) to the contralateral hand (conditioning stimulus).
  PPT will be performed and recorded as descried above prior to and immediately following CPT.
  CPT: Hand will be submerged in an ice bath with the temperature maintained below 3°C for a maximum of 2 minutes. Participants will withdraw their hand when the pain perceived becomes intolerable or 2 minute maximum is reached. Participants will give a numeric pain rating (0-100) at the time of hand removal. Total immersion time (minutes:seconds) and pain rating will be recorded for CPT.
  CPM (primary outcome) will be defined as the absolute numerical difference of PPT after minus before the CPT, with positive values indicating successful pain modulation.
Temporal summation (TS) | Baseline
  Mechanical TS in the present study will be assessed by a wind-up-ratio (WUR) of the volar aspect of the non-dominant arm using a Semmes-Weinstein monofilament (no. 6.45). The perceived intensity of a single stimulus will be compared with that of a series of 10 repetitive stimuli of the same physical intensity. Participants will be asked to give a pain rating for the single stimulus and a pain rating for the series of 10 stimuli as a whole, using a '0-100' numerical rating scale. This procedure will be repeated for three trials, with 1 minute between trials, and performed at different areas of the volar forearm for each trial. The mean pain rating of the 10 series divided by the mean pain rating of the single stimuli will be calculated as WUR. Higher scores indicate greater mechanical TS, indicating an increase in central sensitivity or facilitation.

SECONDARY OUTCOMES:
Central sensitization inventory (CSI) | Baseline
  CSI is a self-report questionnaire indicating the presence of symptoms related to central sensitization syndromes. CSI consists of 25 statements where each statement is evaluated using a 5 point like scale with Never (0), Rarely (1), Sometimes (2), Often (3), and Always (4). This results in a cumulative score of 100. Scores equal to or greater than 40 indicate the likelihood of central sensitization.
Abdominal pain: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a short form | Baseline
  Positive findings for abdominal pain interference, include: mild (50-59), moderate (60-69), or severe (≥70).
Abdominal pain intensity: numeric rating scale | Baseline
  Numeric rating scales recorded for worst, average, and current pain levels, with positive findings as mild (1-4), moderate (5-6), or severe (7-10).
Health-related quality of life (HRQOL) - EQ-5D | Baseline
  The EQ-5D questionnaire descriptive system comprises five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each one with five possible levels: no problems (level 1), slight problems (level 2), moderate problems (level 3), severe problems (level 4), and extreme problems (level 5); as well as a visual analogue scale ranging from 0 to 100 with higher scores indicating 'best health'.
Situational Catastrophizing Questionnaire (SCQ) | Baseline
  SCQ asks participants to reflect on any pain experienced during CPM testing, and to indicate the degree to which they experienced each of 13 thoughts or feelings during this experience, on 5-point Likert scales ranging from (0) not at all to (4) all the time. Total scores range from 0 to 24, with higher score representing greater pain catastrophizing.
Positive and Negative Affective Schedule (PANAS) | Baseline
  This questionnaire includes words describing 10 positive and 10 negative emotions, and requires participants to indicate on a Likert scale (1-5) the extent for which they felt each emotion during the previous week, with higher sub-scores represent greater negative or positive affect styles, respectively.
10-item Perceived Stress Scale (PSS-10) | Baseline
  The PSS-10 evaluates the degree to which individuals believe their life has been unpredictable, uncontrollable, and overloaded during the previous month, using a Likert scale (0-4) for each item, with higher scores representing greater perceived stress.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  Scores for each subscale range from 0 to 21, with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Total comorbidity score | Baseline
  Total comorbidity scores will be calculated as numerical disease counts using health conditions identified on the Self-Administered Comorbidity Questionnaire, a 20-item extraintestinal manifestation (EIM) checklist developed from multiple EIM investigations, and conditions identified on the central sensitization inventory (CSI) (part B). Scores range from 0 to 39 with higher scores indicating greater comorbidity.
MSK pain location | Baseline
  Pain location will be recorded regionally (n=47) using a body diagram. Individuals with generalized pain will be categorically (yes/no) distinguished from those with regional pain using the modified widespread pain criterion which requires having pain in 4 out of 5 pain regions (4 quadrants plus axial pain).
MSK pain - PROMIS Pain Interference 4a | Baseline
  Positive findings for the PROMIS Pain Interference 4a, include: mild (50-59), moderate (60-69), or severe (≥70).
MSK pain intensity - numeric rating scale | Baseline
  Numeric rating scales for pain intensity will be recorded for worst, average, and current pain levels, with positive findings as mild (1-4), moderate (5-6), or severe (7-10)
Health-related quality of life (EQ-5D) | Baseline
  EQ-5D is a standardized instrument for measuring of health-related quality of life. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) each scored on a 5-point Likert scales ranging from (0) no problem to (4) severe. The EQ VAS records the patient's self-rated health on a 0 to 100 vertical visual analogue scale, with higher scores representing better health-related quality of life.
IBD type | Baseline
  IBD subtype recorded from medical charts as Crohn's disease, ulcerative colitis, or unspecified IBD.
IBD duration | Baseline
  Time from initial IBD diagnosis - recorded from medical charts in years.

OTHER OUTCOMES:
Vibration detection threshold (VDT) | Baseline
  VDT will be assessed using a Rydel-Seiffer graded tuning fork (64 Hz, 8/8 scale) placed over bony prominences (styloid process of the ulna and medial malleolus), bilaterally. Participants will verbally indicate the moment they can no longer feel the sensation of vibration, and the value (1-8) will be recorded. VDT of each site will be described as the mean of three trials. Lower scores indicate decreased thresholds and possible peripheral neuropathy.
Semmes-Weinstein monofilament examination (SWME) | Baseline
  SWME of the upper limb will be performed using a 4.56 (4 g) monofilament at six locations divided over the palm and fingers, bilaterally. SWME of the lower limb will be performed using a 5.07 (10 g) monofilament at the pulp of the great toe, as well as the first, third, and fifth metatarsal heads, bilaterally. Participants will confirm (recorded as yes/no) application of the stimulus at each location. Incorrect response at any location indicates possible peripheral neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Siegel, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bliddal H, Danneskiold-Samsoe B. Chronic widespread pain in the spectrum of rheumatological diseases. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):391-402. doi: 10.1016/j.berh.2007.03.005. PMID 17602990
- [Background] Burisch J, Munkholm P. The epidemiology of inflammatory bowel disease. Scand J Gastroenterol. 2015 Aug;50(8):942-51. doi: 10.3109/00365521.2015.1014407. Epub 2015 Feb 17. PMID 25687629
- [Background] M'Koma AE. Inflammatory bowel disease: an expanding global health problem. Clin Med Insights Gastroenterol. 2013 Aug 14;6:33-47. doi: 10.4137/CGast.S12731. eCollection 2013. PMID 24833941
- [Background] Sheth T, Pitchumoni CS, Das KM. Management of Musculoskeletal Manifestations in Inflammatory Bowel Disease. Gastroenterol Res Pract. 2015;2015:387891. doi: 10.1155/2015/387891. Epub 2015 Jun 10. PMID 26170832
- [Background] Zeitz J, Ak M, Muller-Mottet S, Scharl S, Biedermann L, Fournier N, Frei P, Pittet V, Scharl M, Fried M, Rogler G, Vavricka S; Swiss IBD Cohort Study Group. Pain in IBD Patients: Very Frequent and Frequently Insufficiently Taken into Account. PLoS One. 2016 Jun 22;11(6):e0156666. doi: 10.1371/journal.pone.0156666. eCollection 2016. PMID 27332879
- [Background] van Erp SJ, Brakenhoff LK, van Gaalen FA, van den Berg R, Fidder HH, Verspaget HW, Huizinga TW, Veenendaal RA, Wolterbeek R, van der Heijde D, van der Meulen-de Jong AE, Hommes DW. Classifying Back Pain and Peripheral Joint Complaints in Inflammatory Bowel Disease Patients: A Prospective Longitudinal Follow-up Study. J Crohns Colitis. 2016 Feb;10(2):166-75. doi: 10.1093/ecco-jcc/jjv195. Epub 2015 Oct 28. PMID 26512134
- [Background] Palm O, Bernklev T, Moum B, Gran JT. Non-inflammatory joint pain in patients with inflammatory bowel disease is prevalent and has a significant impact on health related quality of life. J Rheumatol. 2005 Sep;32(9):1755-9. PMID 16142874
- [Background] van der Have M, Brakenhoff LK, van Erp SJ, Kaptein AA, Leenders M, Scharloo M, Veenendaal RA, van der Heijde DM, van der Meulen-de Jong AE, Hommes DW, Fidder HH. Back/joint pain, illness perceptions and coping are important predictors of quality of life and work productivity in patients with inflammatory bowel disease: a 12-month longitudinal study. J Crohns Colitis. 2015 Mar;9(3):276-83. doi: 10.1093/ecco-jcc/jju025. Epub 2014 Dec 28. PMID 25547976
- [Background] Brakenhoff LK, van der Heijde DM, Hommes DW. IBD and arthropathies: a practical approach to its diagnosis and management. Gut. 2011 Oct;60(10):1426-35. doi: 10.1136/gut.2010.228866. Epub 2011 May 6. PMID 21551189
- [Background] Levine JS, Burakoff R. Extraintestinal manifestations of inflammatory bowel disease. Gastroenterol Hepatol (N Y). 2011 Apr;7(4):235-41. PMID 21857821
- [Background] Harbord M, Annese V, Vavricka SR, Allez M, Barreiro-de Acosta M, Boberg KM, Burisch J, De Vos M, De Vries AM, Dick AD, Juillerat P, Karlsen TH, Koutroubakis I, Lakatos PL, Orchard T, Papay P, Raine T, Reinshagen M, Thaci D, Tilg H, Carbonnel F; European Crohn's and Colitis Organisation. The First European Evidence-based Consensus on Extra-intestinal Manifestations in Inflammatory Bowel Disease. J Crohns Colitis. 2016 Mar;10(3):239-54. doi: 10.1093/ecco-jcc/jjv213. Epub 2015 Nov 27. No abstract available. PMID 26614685
- [Background] Falling C, Stebbings S, Baxter GD, Gearry RB, Mani R. Profile of musculoskeletal pain in patients with inflammatory bowel disease: a study protocol for assessing the multidimensional experience of self-reported pain. Physical Therapy Reviews. 2018:1-9.
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Curatolo M, Arendt-Nielsen L. Central hypersensitivity in chronic musculoskeletal pain. Phys Med Rehabil Clin N Am. 2015 May;26(2):175-84. doi: 10.1016/j.pmr.2014.12.002. Epub 2015 Feb 4. PMID 25952059
- [Background] Vardeh D, Mannion RJ, Woolf CJ. Toward a Mechanism-Based Approach to Pain Diagnosis. J Pain. 2016 Sep;17(9 Suppl):T50-69. doi: 10.1016/j.jpain.2016.03.001. PMID 27586831
- [Background] Arendt-Nielsen L, Morlion B, Perrot S, Dahan A, Dickenson A, Kress HG, Wells C, Bouhassira D, Drewes AM. Assessment and manifestation of central sensitisation across different chronic pain conditions. Eur J Pain. 2018 Feb;22(2):216-241. doi: 10.1002/ejp.1140. Epub 2017 Nov 5. PMID 29105941
- [Background] Bielefeldt K, Davis B, Binion DG. Pain and inflammatory bowel disease. Inflamm Bowel Dis. 2009 May;15(5):778-88. doi: 10.1002/ibd.20848. PMID 19130619
- [Background] Arendt-Nielsen L, Yarnitsky D. Experimental and clinical applications of quantitative sensory testing applied to skin, muscles and viscera. J Pain. 2009 Jun;10(6):556-72. doi: 10.1016/j.jpain.2009.02.002. Epub 2009 Apr 19. PMID 19380256
- [Background] Sullivan MJ, Thorn B, Haythornthwaite JA, Keefe F, Martin M, Bradley LA, Lefebvre JC. Theoretical perspectives on the relation between catastrophizing and pain. Clin J Pain. 2001 Mar;17(1):52-64. doi: 10.1097/00002508-200103000-00008. PMID 11289089
- [Background] Villemure C, Bushnell CM. Cognitive modulation of pain: how do attention and emotion influence pain processing? Pain. 2002 Feb;95(3):195-199. doi: 10.1016/S0304-3959(02)00007-6. No abstract available. PMID 11839418
- [Background] Boersma K, Linton SJ. How does persistent pain develop? An analysis of the relationship between psychological variables, pain and function across stages of chronicity. Behav Res Ther. 2005 Nov;43(11):1495-507. doi: 10.1016/j.brat.2004.11.006. Epub 2005 Jan 26. PMID 16159591
- [Background] Roth ML, Tripp DA, Harrison MH, Sullivan M, Carson P. Demographic and psychosocial predictors of acute perioperative pain for total knee arthroplasty. Pain Res Manag. 2007 Autumn;12(3):185-94. doi: 10.1155/2007/394960. PMID 17717610
- [Background] Finan PH, Quartana PJ, Smith MT. Positive and negative affect dimensions in chronic knee osteoarthritis: effects on clinical and laboratory pain. Psychosom Med. 2013 Jun;75(5):463-70. doi: 10.1097/PSY.0b013e31828ef1d6. Epub 2013 May 22. PMID 23697467
- [Background] Sterling M, Hodkinson E, Pettiford C, Souvlis T, Curatolo M. Psychologic factors are related to some sensory pain thresholds but not nociceptive flexion reflex threshold in chronic whiplash. Clin J Pain. 2008 Feb;24(2):124-30. doi: 10.1097/AJP.0b013e31815ca293. PMID 18209518
- [Background] Hven L, Frost P, Bonde JP. Evaluation of Pressure Pain Threshold as a Measure of Perceived Stress and High Job Strain. PLoS One. 2017 Jan 4;12(1):e0167257. doi: 10.1371/journal.pone.0167257. eCollection 2017. PMID 28052089
- [Background] Gierthmuhlen J, Enax-Krumova EK, Attal N, Bouhassira D, Cruccu G, Finnerup NB, Haanpaa M, Hansson P, Jensen TS, Freynhagen R, Kennedy JD, Mainka T, Rice ASC, Segerdahl M, Sindrup SH, Serra J, Tolle T, Treede RD, Baron R, Maier C. Who is healthy? Aspects to consider when including healthy volunteers in QST--based studies-a consensus statement by the EUROPAIN and NEUROPAIN consortia. Pain. 2015 Nov;156(11):2203-2211. doi: 10.1097/j.pain.0000000000000227. PMID 26075963
- [Background] Sangha O, Stucki G, Liang MH, Fossel AH, Katz JN. The Self-Administered Comorbidity Questionnaire: a new method to assess comorbidity for clinical and health services research. Arthritis Rheum. 2003 Apr 15;49(2):156-63. doi: 10.1002/art.10993. PMID 12687505
- [Background] Trikudanathan G, Venkatesh PG, Navaneethan U. Diagnosis and therapeutic management of extra-intestinal manifestations of inflammatory bowel disease. Drugs. 2012 Dec 24;72(18):2333-49. doi: 10.2165/11638120-000000000-00000. PMID 23181971
- [Background] Huang V, Mishra R, Thanabalan R, Nguyen GC. Patient awareness of extraintestinal manifestations of inflammatory bowel disease. J Crohns Colitis. 2013 Sep;7(8):e318-24. doi: 10.1016/j.crohns.2012.11.008. Epub 2012 Dec 21. PMID 23265763
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Bernstein CN, Singh S, Graff LA, Walker JR, Miller N, Cheang M. A prospective population-based study of triggers of symptomatic flares in IBD. Am J Gastroenterol. 2010 Sep;105(9):1994-2002. doi: 10.1038/ajg.2010.140. Epub 2010 Apr 6. PMID 20372115
- [Background] Moradkhani A, Beckman LJ, Tabibian JH. Health-related quality of life in inflammatory bowel disease: psychosocial, clinical, socioeconomic, and demographic predictors. J Crohns Colitis. 2013 Jul;7(6):467-73. doi: 10.1016/j.crohns.2012.07.012. Epub 2012 Aug 10. PMID 22884758
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Cohen S, Alper CM, Doyle WJ, Treanor JJ, Turner RB. Positive emotional style predicts resistance to illness after experimental exposure to rhinovirus or influenza a virus. Psychosom Med. 2006 Nov-Dec;68(6):809-15. doi: 10.1097/01.psy.0000245867.92364.3c. Epub 2006 Nov 13. PMID 17101814
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Edwards RR, Smith MT, Stonerock G, Haythornthwaite JA. Pain-related catastrophizing in healthy women is associated with greater temporal summation of and reduced habituation to thermal pain. Clin J Pain. 2006 Oct;22(8):730-7. doi: 10.1097/01.ajp.0000210914.72794.bc. PMID 16988570
- [Background] Buchholz I, Janssen MF, Kohlmann T, Feng YS. A Systematic Review of Studies Comparing the Measurement Properties of the Three-Level and Five-Level Versions of the EQ-5D. Pharmacoeconomics. 2018 Jun;36(6):645-661. doi: 10.1007/s40273-018-0642-5. PMID 29572719
- [Background] Schoepfer AM, Vavricka S, Zahnd-Straumann N, Straumann A, Beglinger C. Monitoring inflammatory bowel disease activity: clinical activity is judged to be more relevant than endoscopic severity or biomarkers. J Crohns Colitis. 2012 May;6(4):412-8. doi: 10.1016/j.crohns.2011.09.008. Epub 2011 Oct 14. PMID 22398068
- [Background] Siegel CA, Whitman CB, Spiegel BMR, Feagan B, Sands B, Loftus EV Jr, Panaccione R, D'Haens G, Bernstein CN, Gearry R, Ng SC, Mantzaris GJ, Sartor B, Silverberg MS, Riddell R, Koutroubakis IE, O'Morain C, Lakatos PL, McGovern DPB, Halfvarson J, Reinisch W, Rogler G, Kruis W, Tysk C, Schreiber S, Danese S, Sandborn W, Griffiths A, Moum B, Gasche C, Pallone F, Travis S, Panes J, Colombel JF, Hanauer S, Peyrin-Biroulet L. Development of an index to define overall disease severity in IBD. Gut. 2018 Feb;67(2):244-254. doi: 10.1136/gutjnl-2016-312648. Epub 2016 Oct 25. PMID 27780886
- [Background] Peyrin-Biroulet L, Panes J, Sandborn WJ, Vermeire S, Danese S, Feagan BG, Colombel JF, Hanauer SB, Rycroft B. Defining Disease Severity in Inflammatory Bowel Diseases: Current and Future Directions. Clin Gastroenterol Hepatol. 2016 Mar;14(3):348-354.e17. doi: 10.1016/j.cgh.2015.06.001. Epub 2015 Jun 11. PMID 26071941
- [Background] Jensen MP, Tome-Pires C, de la Vega R, Galan S, Sole E, Miro J. What Determines Whether a Pain is Rated as Mild, Moderate, or Severe? The Importance of Pain Beliefs and Pain Interference. Clin J Pain. 2017 May;33(5):414-421. doi: 10.1097/AJP.0000000000000429. PMID 27584819
- [Background] Gershon RC, Rothrock N, Hanrahan R, Bass M, Cella D. The use of PROMIS and assessment center to deliver patient-reported outcome measures in clinical research. J Appl Meas. 2010;11(3):304-14. PMID 20847477
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Whitton TL, Johnson RW, Lovell AT. Use of the Rydel-Seiffer graduated tuning fork in the assessment of vibration threshold in postherpetic neuralgia patients and healthy controls. Eur J Pain. 2005 Apr;9(2):167-71. doi: 10.1016/j.ejpain.2004.05.001. PMID 15737809
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Feng Y, Schlosser FJ, Sumpio BE. The Semmes Weinstein monofilament examination as a screening tool for diabetic peripheral neuropathy. J Vasc Surg. 2009 Sep;50(3):675-82, 682.e1. doi: 10.1016/j.jvs.2009.05.017. Epub 2009 Jul 30. PMID 19595541
- [Background] Olaleye D, Perkins BA, Bril V. Evaluation of three screening tests and a risk assessment model for diagnosing peripheral neuropathy in the diabetes clinic. Diabetes Res Clin Pract. 2001 Nov;54(2):115-28. doi: 10.1016/s0168-8227(01)00278-9. PMID 11640995
- [Background] Schreuders TA, Selles RW, van Ginneken BT, Janssen WG, Stam HJ. Sensory evaluation of the hands in patients with Charcot-Marie-Tooth disease using Semmes-Weinstein monofilaments. J Hand Ther. 2008 Jan-Mar;21(1):28-34; quiz 35. doi: 10.1197/j.jht.2007.07.020. PMID 18215749
- [Background] Alqarni AM, Manlapaz D, Baxter D, Tumilty S, Mani R. Test Procedures to Assess Somatosensory Abnormalities in Individuals with Peripheral Joint Pain: A Systematic Review of Psychometric Properties. Pain Pract. 2018 Sep;18(7):895-924. doi: 10.1111/papr.12680. Epub 2018 Mar 6. PMID 29350873
- [Background] Neziri AY, Scaramozzino P, Andersen OK, Dickenson AH, Arendt-Nielsen L, Curatolo M. Reference values of mechanical and thermal pain tests in a pain-free population. Eur J Pain. 2011 Apr;15(4):376-83. doi: 10.1016/j.ejpain.2010.08.011. Epub 2010 Oct 6. PMID 20932788
- [Background] Neziri AY, Limacher A, Juni P, Radanov BP, Andersen OK, Arendt-Nielsen L, Curatolo M. Ranking of tests for pain hypersensitivity according to their discriminative ability in chronic neck pain. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):308-20. doi: 10.1097/AAP.0b013e318295a3ea. PMID 23759706
- [Background] Mlekusch S, Neziri AY, Limacher A, Juni P, Arendt-Nielsen L, Curatolo M. Conditioned Pain Modulation in Patients With Acute and Chronic Low Back Pain. Clin J Pain. 2016 Feb;32(2):116-21. doi: 10.1097/AJP.0000000000000238. PMID 26741741
- [Background] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Background] LeResche L, Turner JA, Saunders K, Shortreed SM, Von Korff M. Psychophysical tests as predictors of back pain chronicity in primary care. J Pain. 2013 Dec;14(12):1663-70. doi: 10.1016/j.jpain.2013.08.008. PMID 24290446
- [Background] Vuilleumier PH, Biurrun Manresa JA, Ghamri Y, Mlekusch S, Siegenthaler A, Arendt-Nielsen L, Curatolo M. Reliability of Quantitative Sensory Tests in a Low Back Pain Population. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):665-73. doi: 10.1097/AAP.0000000000000289. PMID 26222349
- [Background] Meeus M, Roussel NA, Truijen S, Nijs J. Reduced pressure pain thresholds in response to exercise in chronic fatigue syndrome but not in chronic low back pain: an experimental study. J Rehabil Med. 2010 Oct;42(9):884-90. doi: 10.2340/16501977-0595. PMID 20878051
- [Background] Gerhardt A, Eich W, Janke S, Leisner S, Treede RD, Tesarz J. Chronic Widespread Back Pain is Distinct From Chronic Local Back Pain: Evidence From Quantitative Sensory Testing, Pain Drawings, and Psychometrics. Clin J Pain. 2016 Jul;32(7):568-79. doi: 10.1097/AJP.0000000000000300. PMID 26379077
- [Background] Marcuzzi A, Wrigley PJ, Dean CM, Adams R, Hush JM. The long-term reliability of static and dynamic quantitative sensory testing in healthy individuals. Pain. 2017 Jul;158(7):1217-1223. doi: 10.1097/j.pain.0000000000000901. PMID 28328574